CLINICAL TRIAL: NCT06034145
Title: Methacholine Challenge Testing: Comparison of FEV1 and IOS Parameters in Adult Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Allergi- og Lungeklinikken, Elsinore (Network)
Responsible Party: Principal Investigator, Thomas Ringbæk, Principal Investigator, Allergi- og Lungeklinikken, Elsinore
Other Study IDs: Lungeklinikken_Elsinore
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Bronchial Hyperreactivity
Keywords: asthma; oscillometry; spirometry; bronchial hyperreactivity
MeSH Terms: conditions — Bronchial Hyperreactivity; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma: Asthma according to Gina Guidelines
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A classic methacholine challenge test is considered positive when forced expiratory volumen after one second (FEV1) decrease 20%. Impulse oscillometry (IOS) measures airway resistance and reactance, and seems more sensitive to changes in small airways. In adult asthma patients, we compare methacholine challenge test using both FEV1 and IOS.

DETAILED DESCRIPTION:
Asthma is a common chronic disease that is characterized by a history of variable respiratory symptoms and variable expiratory airflow limitation, and usually associated with airway hyperresponsiveness (GINA).

In general, FEV1 is used to test for airway hyperresponsiveness (AHR), and a 20% decrease after methacholine challenge is considered a positive test (Coates 2017; ERJ).

There is increasing recognition that the small airways are involved in 40-80% of patients with asthma, and the function of these airways is overlooked (the "silent zone") when measuring FEV1, which mainly reflects the function of the central airways (Cottini M, J Allergy Clin Immunol Pract 2019; Cottini M, 2022; Postma 2019 Lancet Respir Med).

Small airway dysfunction (SAD) can be assessed by IOS where pressure applied to the airways at a range of frequencies, and components of respiratory resistance and reactance are measured. Resistance at 5 Hz (R5) and 20 Hz (R20), respectively, represent total airway resistance and proximal airway resistance. The difference between these two values can be calculated (R5-R20). High R5-R20 and low reactance at 5 Hz (X5) indicate the presence of SAD.

A recent study showed that patients with a negative methacholine test measured by FEV1 may report asthma-like symptoms and may have a positive test when measured by IOS (Urbankowski; 2021). The question is whether these patients are a subgroup of patients with SAD (based on IOS at baseline) or are characterized in another way.

Knowledge on the proportion of patients with AHR only measured by IOS (not by FEV1) and the characteristics of these patients are sparse.

Hypothesis & Aims The aim of the present study was to determine the proportion of AHR to methacholine measured by FEV1 and IOS, respectively, in patients with diagnosed asthma and to compare patient characteristics and asthma medication in these four groups of patients: 1) negative by FEV1 and IOS; 2) negative by FEV1 but positive by IOS; 3) positive by FEV1 but negative by IOS; 4) positive by both tests.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma (based on symptoms and at least one positive asthma test within the last 5 years (AHR; reversibility to beta2-agonist, ICS, prednisolone; peak flow variation).
* Written informed consent.

Exclusion Criteria:

* patients aged less than 18 years old.
* patients with an exacerbation or lower airway infection within 1 months.
* Pulmonary function test: FEV1 (% pred.) < 60%
* Not able to perform spirometry or body plethysmography.
* Cognitive disorders and not able to answer ACQ.
* Treated with biologics.
* Pregnancy or breastfeeding
* Short-acting beta-agonists 6 h, long-acting beta-agonists 2 days, short-acting anti-muscarinic agent 12 h, Long-acting anti-muscarinic agents 7 days, and Montelukast 3 days before methacholine challenge test (MCT).
* Comorbidity with significant influence on lung function and pulmonary symptoms eg. COPD, bronchiectasis, ischemic heart disease, heart failure, atrial fibrillation, uncontrolled hypertension (>160/100 mmHg), lung cancer, lung resection, BMI>40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional analysis of a single-centered, observational study on adult (≥18 years old) patients referred with known asthma or asthma-like symptoms to a lung specialist clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
ACQ-6 | At entry (Cross sectional)
  Asthma Control Questionnaire (ACQ6) will be used in the 6 sub-score version omitting FEV1 % of predicted
Impulse Oscillometry | At entry
  Resistance at 5Hz (R5), R5-R20, reactance at 5Hz (X5), frequency response (Fres), areal under reactance curve (AX)
Demographic data | At entry
  General demographic data, including age, sex (male/female), body mass index (BMI) (kg/m2), and smoking history will be recorded.
Biomarker | At entry
  Serum eosinophils and hemoglobin will be measured
FeNO | At entry
  Measurement of Exhaled Nitric Oxide by NOBreath
Lung function and body box | At entry
  Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and the percentage of FEV1 in the estimated value will be measured at baseline and after methacholine test by Vyntus, Vyaire Medical. Body plethysmography with residual volumen (RV), total lung capacity (TLC), diffusion capacity of the lungs for carbon monoxide (DLCO), will be measured before methacholine test by Medical Electronic Construction (MEC).
Asthma medication | At entry
  Inhaled corticosteroids (ICS), long-acting beta2agonists (LABA), long-acting muscarinic antagonists (LAMA), Leukotriene antagonist, theophylline, and prednisolone - type and dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ringbæk, MSci, Principal Investigator — Allergy and Lung Clinic Elsinore

IPD SHARING:
Plan to Share IPD: Undecided
Publication in per-reviewed papers;